CLINICAL TRIAL: NCT06458907
Title: A Prospective, Multicenter, Randomized, Clinical Trial of the TricValve Transcatheter Bicaval Valve System in Subjects With Severe Tricuspid Regurgitation (TR).
Brief Title: TRICAV-II Pivotal: TRIcvalve biCAVal Valve System for Severe Tricuspid Regurgitation.
Acronym: TRICAV-II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: P+F Products + Features USA Inc. (Industry)
Collaborators: Meditrial USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-TRIC-005-II
Record Dates: First submitted 2024-06-07; First posted 2024-06-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Disease
Keywords: Tricuspid Regurgitation; Heart Failure
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- TricValve® Device (Device) + Optimal medical therapy (OMT) (Experimental): TricValve® Device (Device) + OMT
  Interventions: Device: TricValve® Transcatheter Bicaval Valve System; Drug: Optimal medical therapy
- Optimal medical therapy (OMT) Alone (Active Comparator): OMT can prevent heart attacks and heart failure with medications like blood thinners, cholesterol drugs, and blood pressure meds.
  Interventions: Drug: Optimal medical therapy
- TricValve Single Arm Registry (Experimental): Patients who fulfil any of the screening criteria to participate in a parallel singe-arm registry.
  Interventions: Device: TricValve® Transcatheter Bicaval Valve System; Drug: Optimal medical therapy

INTERVENTIONS:
Device: TricValve® Transcatheter Bicaval Valve System — TricValve® Device (Device) Group subjects will undergo TricValve® implantation and will continue to be managed with optimal medical therapies.
  Other Names: TricValve System
  Arms: TricValve Single Arm Registry; TricValve® Device (Device) + Optimal medical therapy (OMT)
Drug: Optimal medical therapy — Optimal medical therapy
  Other Names: OMT

SUMMARY:
The Investigational Device is the TricValve Transcatheter Bicaval Valve System (also referred to as the TricValve System).

The bioprosthesis is available in two different diameters for each model (SVC and IVC) specifically designed to adapt to the anatomic features of the superior vena cava (SVC) and inferior vena cava (IVC).

The SVC and IVC valves are single use, sterile devices provided in two sizes each, for a total of four valve sizes. The valves are designed for heterotopic caval implantation without perturbing the native tricuspid valve. The valves are made of bovine pericardium leaflets sutured on a nitinol self-expanding stent system.

The SVC and IVC valves are provided pre-mounted in two separate TricValve Delivery Systems, and are individually packaged into two separate boxes, provided sterile and ready to use. The two TricValve Delivery Systems deliver the two valves percutaneously into the SVC and IVC via femoral vein access using a transvenous approach.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized controlled pivotal clinical trial to evaluate the safety and effectiveness of the TricValve System with Optimal Medical Therapy (OMT) compared to OMT alone in the treatment of patients with severe TR and caval reflux (CR).

The TricValve System received Breakthrough Device Designation from the US FDA.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be 18 years or older.
2. Severe tricuspid regurgitation (TR), as determined by Echo Core Lab.
3. NYHA Class III-IVa or heart failure (HF) admission in the past 6 months.
4. Subject is treated with stable OMT for at least 30 days.
5. The local Heart Team and Independent Eligibility Committee (IEC) determine that the patient is eligible
6. For females of childbearing potential, negative pregnancy test.
7. Capable and willing to provide signed informed consent.

Exclusion Criteria:

1. Recent Myocardial Infarction (MI), stroke or Cerebrovascular Accident (CVA); major cardiovascular surgery within 90 days.
2. Subject requires another planned major cardiac procedure.
3. Left Ventricular Ejection Fraction (LVEF) ≤ 30% on echocardiography.
4. Evidence of intracardiac, inferior vena cava (IVC), or femoral venous mass, thrombus or vegetation.
5. Tricuspid stenosis.
6. Severe right ventricular dysfunction.
7. Cardiac amyloidosis.
8. Pulmonary artery systolic pressure (PASP) >65 mmHg.
9. Lower extremity venous thrombosis and/or the presence of an IVC filter at the time of or 6 months prior to TricValve procedure.
10. Hemodynamically significant pericardial effusion.
11. Patient with refractory heart failure requiring advanced intervention
12. Any known allergy or hypersensitivity to nitinol, bovine tissue or contrast media that cannot be adequately treated with pre-medication.
13. Unable to tolerate anticoagulation/antiplatelet therapy.
14. Hemodynamic instability, cardiogenic shock, inotropic support, intra-aortic balloon pump or acute heart failure within 30 days prior to the TricValve procedure.
15. Life expectancy lower than 12 months.
16. Platelet count < 75,000/mm3.
17. Child-Pugh Severity Class C (10-15 points).
18. Severe renal insufficiency with Estimated Glomerular Filtration Rate (eGFR) ≤ 25 mL/min/1.73 m2 or dialysis.
19. Endocarditis or active/ongoing infection requiring antibiotics.
20. Unable to walk at least 60 meters in a 6minute walk test.
21. Known bleeding or clotting disorders or patient refuses blood transfusion.
22. Active gastrointestinal (GI) bleeding within 3 months of TricValve procedure.
23. Presence of significant congenital heart disease including but not limited to hemodynamically significant atrial septal defect, Right ventricular (RV) dysplasia, and arrhythmogenic RV.
24. Participation in other investigational devices or drug study.
25. Any other condition that would preclude ability to meet study requirements in the opinion of the investigator.
26. Psychiatric/behavioral issues or other medical or social conditions that preclude valid consent and follow-up.
27. Pregnant or breastfeeding subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 Month, 12 Months
  Number of Cardiovascular Deaths at 30 Days.
Q-wave myocardial infarctions | 1 Month
  Number of myocardial infarctions at 30 Days.
Disabling stroke | 1 Month
  Number of days until death.
Life threatening bleeding | 1 Month
  Number of days until death.
Pulmonary embolism | 1 Month
  Number of days until death.
Renal failure requiring dialysis | 1 Month
  Number of days until new renal replacement therapy.
Major access-site, vascular, or cardiac structural complications | 1 Month
  Number of days until death.
Emergency surgery or intervention related to the device/procedure complications | 1 Month
  Number of days until emergency surgery or intervention.
Reduction in Caval Reflux (CR) | 6 Months
  Reduction in CR, measured by echocardiography
Kansas City Cardiomyopathy Questionnaire (KCCQ Score) | 6 Months, 12 Months
  Change in KCCQ score (score ranges between 0 and 100)
New York Heart Association (NYHA Class) | 6 Months, 12 Months
  Change in NYHA class (range from I to IV)
Six Minute Walking Test (6MWT) | 6 Months, 12 Months
  Change in walking distance
Right Ventricular Assist Device (RVAD) implantation or heart transplant | 12 Months
  Number of days until Right Ventricular Assist Device (RVAD) implantation or heart transplant
Tricuspid valve surgery or percutaneous tricuspid intervention | 12 Months
  Number of days until tricuspid valve surgery or percutaneous tricuspid intervention
Heart Failure Events | 12 Months
  Number of heart failure episodes including hospitalization, or worsening heart failure

SECONDARY OUTCOMES:
Secondary Safety Endpoint (measured at 1 year) | 12 Months
  The percentage of subjects with Device- and/or Procedure-related MAEs through 1 year.
All-Cause mortality | 3 Months, 6 Months, and 12 Months
  Number of days until death.
Kansas City Cardiomyopathy Questionnaire (KCCQ Score) | 3 Months, 6 Months, and 12 Months
  Change in KCCQ score (score ranges between 0 and 100)
Right Ventricular Assist Device (RVAD) implantation or heart transplant | 3 Months, 6 Months, and 12 Months
  Number of days until Right Ventricular Assist Device (RVAD) implantation or heart transplant.
Six Minute Walking Test (6MWT) | 3 Months, 6 Months, and 12 Months
  Change in walking distance
Atrial Fibrillation | 3 Months, 6 Months, and 12 Months
  Days to new onset of atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Scripps Memorial Hospital La Jolla, San Diego, California
  - Tampa General Hospital, Tampa, Florida
  - Northshore Evanston Hospital, Evanston, Illinois
  - Ascension Medical Group St. Vincent The Heart Center of Indiana, Indianapolis, Indiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Columbia University Medical Center/ NewYork Presbyterian Hospital, Irving, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Pinnacle, Harrisburg, Pennsylvania
  - Houston Methodist, Houston, Texas
  - University of Texas (Memorial Hermann), Houston, Texas
  - Intermountain Heart Institute - Intermountain Medical Center, Murray, Utah
  - MedStar Washington Hospital Center, Multiple Locations, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amat-Santos IJ, Estevez-Loureiro R, Sanchez-Recalde A, Cruz-Gonzalez I, Pascual I, Mascherbauer J, Abdul-Jawad Altisent O, Nombela-Franco L, Pan M, Trillo R, Moreno R, Delle Karth G, Blasco-Turrion S, Sanchez-Luna JP, Revilla-Orodoea A, Redondo A, Zamorano JL, Puri R, Iniguez-Romo A, San Roman A. Right heart remodelling after bicaval TricValve implantation in patients with severe tricuspid regurgitation. EuroIntervention. 2023 Aug 7;19(5):e450-e452. doi: 10.4244/EIJ-D-23-00077. No abstract available. PMID 37083622
- [Result] Blasco-Turrion S, Briedis K, Estevez-Loureiro R, Sanchez-Recalde A, Cruz-Gonzalez I, Pascual I, Mascherbauer J, Abdul-Jawad Altisent O, Nombela-Franco L, Pan M, Trillo R, Moreno R, Delle Karth G, Sanchez-Luna JP, Gonzalez-Gutierrez JC, Revilla-Orodoea A, Zamorano JL, Gomez-Salvador I, Puri R, San Roman JA, Amat-Santos IJ. Bicaval TricValve Implantation in Patients With Severe Symptomatic Tricuspid Regurgitation: 1-Year Follow-Up Outcomes. JACC Cardiovasc Interv. 2024 Jan 8;17(1):60-72. doi: 10.1016/j.jcin.2023.10.043. Epub 2023 Dec 6. PMID 38069986
- See also: Products & Features, manufacturer of TricValve® Transcatheter Bicaval Valve System — https://productsandfeatures.com/
- See also: Meditrial Clinical Research Organization — http://www.meditrial.net